CLINICAL TRIAL: NCT07073859
Title: Fluid Responsiveness Assessment in Pediatric Intensive Care Units: a Nationwide Clinical Practice Analysis
Brief Title: Fluid Responsiveness Assessment in Children
Acronym: FRAICHE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/94; CER-BDX 2024 - 31 (Other: Comité d'Ethique de la Recherche du Centre Ethique et Recherche en Santé de Bordeaux)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Circulatory Failure; Shock State
Keywords: Circulatory failure; Fluid therapy; Fluid responsiveness; Critical care
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluid expansion — Data will be collected retrospectively, after fluid expansion administration, by the prescribing physician through. These data will be collected from standard monitoring and/or from the patient's medical record. Data will therefore only be collected at a single point in time.

SUMMARY:
Fluid responsiveness assessment is a major issue in intensive care. Since fewer fluid responsiveness tests can be used children, fluid expansion prescriptions are often based on professional practices due to the absence of guidelines. This observational, cross-sectional, multicentric study is an evaluation of professional practices regarding fluid expansions in pediatric intensive care units. The main objective will be to describe the proportion of fluid expansions that are administered following an assessment of fluid responsiveness.

DETAILED DESCRIPTION:
Fluid expansion is the cornerstone of acute circulatory failure treatment. Although this therapy drastically reduced mortality, several studies in recent years have highlighted the adverse effects of excessive fluid expansion (leading to fluid overload). Currently, the search for indicators to predict fluid responsiveness is a major issue in intensive care units (ICU). These indicators are based on Franck-Starling's law: if small changes in preload lead to an increase in cardiac output, then fluid responsiveness can be expected. This assessment is necessary but must be as simple as possible in an emergency setting such as ICU. Although several fluid responsiveness tests are available in adults, they are underused in current practice. In children, the only validated indicator (respiratory variability of peak aortic velocity) can only be used in the absence of any spontaneous respiratory movement, a rare situation in practice. Thus, fluid expansion prescriptions in pediatric ICU (PICU) are based on professional practices that are often heterogeneous due to the absence of evidence-based guidelines. An evaluation of professional practices is a first step towards standardizing practices.

This study is an evaluation of professional practices regarding fluid expansion in PICU. The main objective will be to describe the proportion of fluid expansions that are administered following an assessment of fluid responsiveness.

We will conduct an observational, cross-sectional, multicentric study in French PICU. Data will be collected retrospectively, after fluid expansion administration, by the prescribing physician through a electronic CRF (RedCAP). These data will be collected from standard monitoring and/or from the patient's medical record. Data will therefore only be collected at a single point in time.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 15 years old
* Hospitalization in a pediatric intensive care unit
* Prescription by the attending physician of a fluid expansion in order to increase cardiac output and restore the patient's circulatory function, which the physician has judged to be impaired. Fluid expansion is defined as a rapid intravenous infusion (<30min) of a high volume (>10ml/kg or 250ml) of an isotonic crystalloid solution, albumin, or fresh frozen plasma. The decision to administer a fluid expansion and the type of fluid administered are left to the discretion of the physician (current practice).

Exclusion Criteria:

* Patient less than 37 weeks' corrected gestational age
* Univentricular circulatory physiology
* Mechanical circulatory support
* Opposition of the patient or his/her parents or legal guardians to data collection

Ages: 37 Weeks to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fluid expansion prescriptions in pediatric ICU (PICU)
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Percentage of fluid expansions preceded by a fluid responsiveness assessment | Day 0
  It will be collected by auditing the prescribing physician after each fluid expansion administration.

SECONDARY OUTCOMES:
Percentage of each fluid responsiveness test used | Day 0
Percentage of fluid responsiveness tests used with all of the validity criteria | Day 0
Mean volume of fluid expansions | Day 0
Mean duration of fluid expansions | Day 0
Percentage of fluid expansion efficacy evaluations based on cardiac output measurement | Day 0
Association between fluid responsiveness assessment and prescribing physician's seniority | Day 0
Association between fluid responsiveness assessment and prescribing physician's specialty | Day 0
Association between fluid responsiveness assessment and patient's age | Day 0
Association between fluid responsiveness assessment and origin of hemodynamic failure | Day 0
Association between fluid responsiveness assessment and history of previous fluid expansion | Day 0
Association between fluid responsiveness assessment and inotropic or vasopressor support | Day 0
Association between fluid responsiveness assessment and strict criteria for acute circulatory failure | Day 0
Association between fluid responsiveness assessment and volume of fluid expansion | Day 0
Association between fluid responsiveness assessment and fluid administered. | Day 0

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Site Sud - CHU d'Amiens Picardie, Amiens, France
  - CHU d'Angers, Angers, France
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux, France
  - Hôpital Morvan - CHU de Brest, Brest, France
  - Hôpital Louis Pradel - Hospices Civils de Lyon, Bron, France
  - CHU Caen Normandie, Caen, France
  - Site Estaing - CHU de Clermont-Ferrand, Clermont-Ferrand, France
  - Hôpital d'Enfants - CHU de Dijon-Bourgogne, Dijon, France
  - Hôpital Raymond Poincaré - Assistance Publique - Hôpitaux de Paris, Garches, France
  - Hôpital Couple-Enfant -Hôpital Couple-Enfant, Grenoble, France
  - Hôpital Felix Guyon (Saint Denis) - CHU de la Réunion, La Réunion, France
  - Hôpital Kremlin Bicêtre - Assistance Publique - Hôpitaux de Paris, Le Kremlin-Bicêtre, France
  - Hôpital Marie-Lannelongue, Le Plessis-Robinson, France
  - Hôpital Jeanne de Flandre - CHRU de Lille, Lille, France
  - Hôpital de la mère et de l'enfant - CHU de Limoges, Limoges, France
  - Hôpital de la Timone - Assistance Publique - Hôpitaux de Marseille, Marseille, France
  - Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier, France
  - Hôpital mère-enfant - CHU de Nantes, Nantes, France
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France
  - Hôpital Trousseau - Assistance Publique - Hôpitaux de Paris, Paris, France
  - Hôpital Necker-Enfants Malades - Assistance Publique - Hôpitaux de Paris, Paris, France
  - Hôpital Robert Debré - Assistance Publique - Hôpitaux de Paris, Paris, France
  - CHU de Bordeaux - Hôpital Cardiologique Haut-Lévêque, Pessac, France
  - La Milétrie - CHU de Poitiers, Poitiers, France
  - Hôpital d'enfants - American Memorial Hospital - CHU de Reims, Reims, France
  - Hôpital Sud - CHU de Rennes, Rennes, France
  - Hôpital Charles-Nicolle - CHU de Rouen, Rouen, France
  - Hôpital de Hautepierre - Hôpitaux Universitaires de Strasbourg, Strasbourg, France
  - Hôpital des enfants - Hôpital des enfants, Toulouse, France
  - Hôpital Clocheville - CHRU de Tours, Tours, France
  - Hôpitaux de Brabois - CHRU de Nancy, Vandœuvre-lès-Nancy, France